CLINICAL TRIAL: NCT02244801
Title: Donor-Alloantigen-Reactive Regulatory T Cell (darTreg) Therapy in Renal Transplantation: A ONE Study Clinical Trial
Brief Title: Donor-Alloantigen-Reactive Regulatory T Cell (darTreg) Therapy in Renal Transplantation (The ONE Study )
Acronym: DART
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Principal Investigator, Sang-Mo Kang, Associate Professor of Surgery, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONEdarTreg14
Record Dates: First submitted 2014-09-11; First posted 2014-09-19 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Other): 3 subjects treated with a target dose of 300 million darTreg with the possibility of expanding to 5 patients if safety signals should require additional patients be observed at the 300 million dose.
  The first subject in each dosing cohort will be monitored for 4 weeks after darTreg infusion. Following the 4 week observation period, the study team will conduct a thorough review of all available data to ensure that there are no safety signals and to make a determination about proceeding with additional patients.
  Interventions: Drug: darTreg infusion
- Cohort 2 (Other): The second cohort will comprise a minimum of 3 and up to 5 subjects treated at a target dose of 900 million darTreg, depending on how many patients were required to be treated in lower dose group.
  The first subject in each dosing cohort will be monitored for 4 weeks after darTreg infusion. Following the 4 week observation period, the study team will conduct a thorough review of all available data to ensure that there are no safety signals and to make a determination about proceeding with additional patients.
  Interventions: Drug: darTreg infusion

INTERVENTIONS:
Drug: darTreg infusion — The first subject in each dosing cohort will be monitored for 4 weeks after darTreg infusion. Following the 4 week observation period, the study team will conduct a thorough review of all available data to ensure that there are no safety signals and to make a determination about proceeding with additional patients. sBc production for darTreg manufacturing for the second subject in each cohort may be initiated but the second subject may not undergo leukapheresis until the safety review is complete.
  Once the last subject in the first cohort reaches week 4 post-infusion, the DSMB will conduct a thorough review of all available data to make a determination about proceeding with additional patients at the lower dose or proceeding to the second dosing cohort. sBc production for darTreg manufacturing for the subsequent subject may be initiated but the patient may not undergo leukapheresis until the DSMB( Data Safety and Monitoring Board ) has approved enrollment of subsequent subjects.
  Other Names: darTregs

SUMMARY:
This Phase I pilot study will evaluate the safety, and tolerability of darTreg infusion for adult, de novo, living donor renal transplant recipients.

DETAILED DESCRIPTION:
A single-center, open-label, dose-escalation pilot trial of a single infusion of darTregs in two dosing cohorts. This study is an independent single-center clinical trial. However, the organizational and mechanistic infrastructure of the study will be provided by the ONE Study project, a European Union funded collaborative project, whose objective is to assess distinct purified hematopoietic immunoregulatory cells as clinical therapies in solid organ transplantation. This study is one of multiple clinical trials within the framework of The ONE Study project, based on the same general design.

ELIGIBILITY:
Inclusion Criteria: (organ donor eligibility)

1. Eligible for live kidney donation
2. At least 18 years of age
3. An ABO blood type compatible with the organ recipient
4. Willing and able to provide a blood sample for The ONE Study IM (Immune Monitoring) Subproject
5. Willing to provide personal and medical/biological data for the trial analysis
6. Eligible to give blood for B cell source prior to organ donation
7. Signed and dated written informed consent*. *For subjects unable to read and/or write, oral informed consent observed by an independent witness is acceptable if the subject has fully understood oral information given by the Investigator. The witness should sign the consent form on behalf of the subject.

In signing the donor information sheet/informed consent form (DIS/ICF), organ donors agree to undergo phlebotomy to provide donor B cells for the production of darTreg, to provide a blood sample for the IM Subproject, and permit access to their medical records for the collection of specified demographic and medical/biological data for the trial.

Organ Recipient eligibility:

A prospective kidney transplant recipient is eligible for enrollment into the study if all of the following inclusion criteria apply:

1. Chronic renal insufficiency necessitating kidney transplantation and approved to receive a primary kidney allograft from a living donor
2. At least 18 years of age
3. Able to commence the immunosuppressive regimen at the protocol-specified time point
4. Willing and able to participate in The ONE Study IM and HEC (Health-Economics Subproject) subprojects
5. Adequate venous access to support leukapheresis
6. Signed and dated written informed consent*.

   * For patients unable to read and/or write, oral informed consent observed by an independent witness is acceptable if the patient has fully understood oral information given by the Investigator. The witness should sign the consent form on behalf of the patient.

Exclusion Criteria: (organ donor)

If a prospective donor fulfills any of the following criteria, they are ineligible for the trial:

1. Genetically identical to the prospective organ recipient at the HLA (human leukocyte antigen) loci (0-0-0 mismatch)
2. CMV-positive and donating to a CMV-negative recipient
3. Exposure to any investigational agents at the time of kidney donation, or within 28 days prior to kidney donation
4. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
5. Subjects unable to freely give their informed consent (e.g. individuals under legal guardianship).

Exclusion criteria (organ recipient)

1. Patient has previously received any tissue or organ transplant other than the planned kidney graft
2. Known contraindication to the protocol-specified treatments / medications
3. Genetically identical to the prospective organ donor at the HLA (human leukocyte antigen) loci (0-0-0 mismatch)
4. PRA (panel reactive antibody) grade > 40% within 6 months prior to enrollment
5. Previous treatment with any desensitization procedure (with or without IVIg)
6. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non-metastatic basal/squamous cell carcinoma of the skin)
7. Evidence of significant local or systemic infection
8. HIV-positive, EBV-negative or suffering chronic viral hepatitis
9. CMV-negative and receiving a kidney from a CMV-positive donor
10. Significant liver disease, defined as persistently elevated AST (aspartate aminotransferase) and/or ALT(alanine aminotransferase) levels > 2 x ULN (Upper Limit of Normal range)
11. Malignant or pre-malignant hematological conditions
12. Neutrophils < 1000/μl ; platelets < 100,000/μl
13. Regulatory T cells present in peripheral blood at <30/µL
14. Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives
15. Any condition which, in the judgment of the Investigator, would place the subject at undue risk
16. Ongoing treatment with systemic immunosuppressive drugs at study entry
17. Patients who have received anti-T cell therapy within 30 days prior to transplant surgery
18. Participation in another clinical trial during the study or within 28 days prior to planned study entry
19. Female patients of reproductive potential with a positive pregnancy test at enrollment
20. Female patients who are breast-feeding
21. All female patients of reproductive potential* UNLESS the patient is willing to use an acceptable birth control for the duration of the study unless the patient chooses abstinence (she chooses to avoid heterosexual intercourse completely) (See Table 2. Acceptable Contraception Methods for Females of Reproductive Potential)
22. Male patients unwilling to use a reliable and effective form of contraception for 3 months after darTreg dosing
23. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule
24. Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel
25. Patients unable to freely give their informed consent (e.g. individuals under legal guardianship).

    * Females of reproductive potential include girls who have entered puberty and all women who have a uterus and have not passed through menopause. Menopause is the permanent end of menstruation and fertility. Menopause should be clinically confirmed by a patient's healthcare practitioner. Some commonly used diagnostic criteria include 1) 12 months of spontaneous amenorrhea (not amenorrhea induced by a medical condition or medical therapy) or 2) postsurgical from a bilateral oophorectomy.

Exclusion Criteria B (organ recipient)

Below are exclusion criteria to be assessed post-transplantation and prior to darTreg infusion. Subjects who meet any of these criteria should not receive a darTreg-infusion:

1. Unacceptable darTreg product.
2. Delayed graft function (requiring dialysis post-transplant).
3. Requiring oxygen supplementation to keep capillary oxygen saturations >95%.
4. Any medical or technical complications (e.g. myocardial infarction, urine leak, wound dehiscence, pneumonia, ongoing fevers, etc.) that in the judgment of the investigators or responsible clinician would put the subject at undue risk.-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection (BCAR) following renal transplantation. | 60 weeks post renal transplantation
  Explore the immunomodulatory potential, safety and tolerability of a single infusion of darTregs as adjunct immunosuppressive treatment through the incidence of biopsy-confirmed acute rejection (BCAR) within 60 weeks following renal transplantation.

SECONDARY OUTCOMES:
Time to first acute rejection episode | 60 weeks post renal transplantation
Severity of acute rejection episodes | 60 weeks post renal transplantation
  severity of acute rejection episodes based on response to treatment and histological scoring
Total immunosuppressive burden at 60 weeks post-transplantation | 60 weeks post renal transplantation
  Total immunosuppressive burden assessed at last study visit
Prevention of chronic graft dysfunction (chronic rejection or IF/TA) | 60 weeks post renal transplantation
  chronic graft dysfunction assessed by clinical (impairment of GFR) and histopathological (Banff staging) measures
Incidence of post-transplant dialysis, inclusion on the transplant waiting list or re-transplantation following graft loss through rejection | 60 weeks post renal transplantation
Avoidance of drug-related complications by immunosuppressant reduction | 60 weeks post renal transplantation
  Assessed by the incidence of reported adverse drug reactions
Biochemical disturbances caused by cell infusion | 1 week
  Assessed by Incidence of acute toxicities associated with infusion of the cell product
Over-suppression of the immune system assessed by the incidence of major and/or opportunistic infections especially CMV (cytomegalovirus ), EBV (Epstein-Barr virus) and polyoma virus | 60 weeks post renal transplantation
Incidence of neoplasia | 60 weeks post renal transplantation
Incidence of patients treated for subclinical acute rejection | 60 weeks post transplantation

OTHER OUTCOMES:
Incidence of malignancies arising directly from darTreg infusion | 60 weeks
incidence of autoimmune disorders | 60 weeks post transplantation
A Health-Economics Subproject will evaluate the health-related qualify-of-life of trail patients using patient-reported outcome measures | 60 weeks post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Mo Kang, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco - Transplant Department. 513 Parnassus Ave HSE 504, San Francisco, California, United States

REFERENCES:
- [Background] ICH Harmonised Tripartite Guideline. Statistical principles for clinical trials. International Conference on Harmonisation E9 Expert Working Group. Stat Med. 1999 Aug 15;18(15):1905-42. No abstract available. PMID 10532877
- [Background] Francillon A, Pickering G, Belorgey C. Exploratory clinical trials: implementation modes & guidelines, scope and regulatory framework. Therapie. 2009 May-Jun;64(3):149-59. doi: 10.2515/therapie/2009022. Epub 2009 Aug 13. English, French. PMID 19671427
- [Background] Morris PJ. Transplantation--a medical miracle of the 20th century. N Engl J Med. 2004 Dec 23;351(26):2678-80. doi: 10.1056/NEJMp048256. No abstract available. PMID 15616201
- [Background] Sayegh MH, Carpenter CB. Transplantation 50 years later--progress, challenges, and promises. N Engl J Med. 2004 Dec 23;351(26):2761-6. doi: 10.1056/NEJMon043418. No abstract available. PMID 15616214
- [Background] Gibson T, Medawar PB. The fate of skin homografts in man. J Anat. 1943 Jul;77(Pt 4):299-310.4. No abstract available. PMID 17104936
- [Background] Medawar PB. The behaviour and fate of skin autografts and skin homografts in rabbits: A report to the War Wounds Committee of the Medical Research Council. J Anat. 1944 Oct;78(Pt 5):176-99. No abstract available. PMID 17104960
- [Background] Halloran PF. Immunosuppressive drugs for kidney transplantation. N Engl J Med. 2004 Dec 23;351(26):2715-29. doi: 10.1056/NEJMra033540. No abstract available. PMID 15616206
- [Result] MERRILL JP, MURRAY JE, HARRISON JH, GUILD WR. Successful homotransplantation of the human kidney between identical twins. J Am Med Assoc. 1956 Jan 28;160(4):277-82. doi: 10.1001/jama.1956.02960390027008. No abstract available. PMID 13278189
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407